CLINICAL TRIAL: NCT00761943
Title: "Adhesive Capsulitis-Correlating Clinical Disease State With Color Doppler Ultrasound"
Brief Title: Correlating Clinical Disease State With Color Doppler Ultrasound
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Rosemary A. Sanders, Research Coordinator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 061180
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Bursitis; Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We are trying to see if ultrasound is a good tool for looking at the changes that happen on the inside of the shoulder due frozen shoulder.

DETAILED DESCRIPTION:
Disease Prevalence:

Orthopaedic surgeons are frequently asked to evaluate patients with stiff and painful shoulders. Among the most common causes for such clinical condition is adhesive capsulitis (or frozen shoulder), which is thought to affect approximately 2-5% of the general population. The incidence in patients with diabetes is much higher, up to 29% in some studies.

Clinical Summary of Adhesive Capsulitis:

Adhesive Capsulitis may be summarized briefly as the clinical syndrome of shoulder pain and progressive loss of motion and eventual improvement of symptoms. The cause is classified as either primary (idiopathic) or secondary, if due to a known precipitating condition. Risk factors associated with developing adhesive capsulitis include diabetes, female sex, middle to older age, and thyroid disease. Secondary causes of adhesive capsulitis include trauma, shoulder surgery, degenerative arthritis, rotator cuff tears, or prolonged immobilization.

The condition is characterized functionally by loss of both active and passive range of motion and anatomically by thickening and contracture of the joint capsule. The term "Adhesive Capsulitis" was coined by Neviaser when he noted the contracted capsule peeled from the humeral head like "adhesive plaster from skin". A broader term "Frozen Shoulder" was used by Codman in 1934 to describe this and related conditions. There is a commonly accepted progression of three clinical phases: painful freezing, stiff/frozen phase, and eventually thawing with slow return of motion. Many patients will have some residual loss of motion for several years. For people with diabetes, residual, permanent loss of motion can be as much as 50%. The natural history of the disease has been shown to be more dismal than once thought.

Pathology of the Disease:

Histopathologic changes that occur in the joint capsule and synovial lining are cellular changes of chronic inflammation, fibrosis, perivascular infiltration in the subsynovial layer and increased vascularity. There is some debate as to whether the disease is primarily inflammatory or fibrotic in nature and there is support for both, depending on the stage of disease. Some have shown that arthroscopy reveals a highly vascular, red, inflamed synovium. Neviaser defined four stages of arthroscopic adhesive capsulitis ranging from acute synovitis to chronic adhesions. The pathology is not clearly understood and this makes optimal treatment more difficult to determine.

Limitations of Current Imaging Studies:

Imaging modalities commonly used to evaluate the shoulder such as x-ray (to rule out arthritic changes or fractures) are unremarkable in primary adhesive capsulitis. Traditional arthrograms or contrast Magnetic Resonance Imaging may show decreased capsular volume and edema but are invasive and expensive tests. Magnetic Resonance Arthrogram shows thickening of the coracohumeral ligament and the joint capsule in the area of the rotator interval. Although MRI can demonstrate edema and inflammatory changes, its cost seems prohibitive to follow clinical disease on a serial basis, perhaps monthly as the disease progresses. Ultrasound is a much more likely candidate for serial examination.

Successful Use of Ultrasound in Rheumatoid Wrist Studies:

Recent reports in the literature have shown color doppler ultrasound (CDUS) to be a promising tool for estimation of synovial inflammatory activity in rheumatoid arthritis. Researchers used specific quantitative criteria to measure the resistivity index of small blood vessels in the synovium and color pixel fraction. Both measures attempt to quantify vascularity as a surrogate indicator of inflammation in the joint capsule. In a subsequent study they injected the wrists with corticosteroid and then obtained ultrasound images one month later which showed changes in the resistivity index and color pixel fraction that correlated with the improved clinical evaluation and functional improvements.

Ultrasound in Adhesive Capsulitis:

Ultrasound study of the shoulder has many benefits over MRI/MRA including: no contraindications or risk to patients, non-invasive, and relatively low cos. Ultrasound is comparable to MRI in studying the synovium with much less downside. Despite is theoretical advantages; there are limited studies in the literature reporting on color doppler ultrasound to evaluate adhesive capsulitis of the shoulder. In one study, researchers correlated ultrasound findings with arthroscopic findings and concluded that ultrasound can provide an early, accurate diagnosis of adhesive capsulitis. Their criteria, however, were qualitative using echotexture and increased doppler flow to indicate increased vascularity. No quantitative measurements were made.

Clinical Importance of Proposed Study:

Although the objective in treating patients with adhesive capsulitis is clear (to restore full, pain-free motion and unrestricted shoulder function) the optimal treatment remains unclear. This is due in part because there is no clear consensus on diagnosis, poor understanding of the pathology, and difficulty comparing the effectiveness of treatment regimens. As in many poorly defined medical conditions, multiple, different empiric treatments are employed with varying success. If we could more clearly identify diagnostic criteria and reproducibly stage the disease we could then more reliably and scientifically compare treatment approaches and thus provide a real benefit to many patients with this common condition. Our proposed study is an important step in this process.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18 to 80.
* Clinical diagnosis of Adhesive Capsulitis of the shoulder.

Exclusion Criteria:

* Previous shoulder surgery.
* Secondary Adhesive Capsulitis related to trauma, surgery or other known causes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 80 with Adhesive Capsulitis of the shoulder without previous shoulder surgery. Not including patients with secondary adhesive capsulitis related to trauma, surgery or other known cause.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To use color doppler ultrasound to grade inflammatory changes in the rotator interval of patients with adhesive capsulitis. | Patients will be evaluated at each of their regularly scheduled clinic follow-up visits.

SECONDARY OUTCOMES:
To use color doppler ultrasound to quantitatively measure inflammation of the joint capsule in subjects with adhesive capsulitis. Specific metrics that measure vascularity as a surrogate for inflammation will be used. | Patients will be evaluated at each of their regularly scheduled clinic follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Warren R. Dunn, M.D., Principal Investigator — Vanderbilt Orthopaedics and Rehabilitation
Locations (1):
- Vanderbilt Orthopaedics and Rehabilitation, Nashville, Tennessee, United States

REFERENCES:
- [Background] Balci N, Balci MK, Tuzuner S. Shoulder adhesive capsulitis and shoulder range of motion in type II diabetes mellitus: association with diabetic complications. J Diabetes Complications. 1999 May-Jun;13(3):135-40. doi: 10.1016/s1056-8727(99)00037-9. PMID 10509873
- [Background] Dias R, Cutts S, Massoud S. Frozen shoulder. BMJ. 2005 Dec 17;331(7530):1453-6. doi: 10.1136/bmj.331.7530.1453. PMID 16356983
- [Background] Hannafin JA, Chiaia TA. Adhesive capsulitis. A treatment approach. Clin Orthop Relat Res. 2000 Mar;(372):95-109. PMID 10738419
- [Background] Kordella T. Frozen shoulder & diabetes. Frozen shoulder affects 20 percent of people with diabetes. Proper treatment can help you work through it. Diabetes Forecast. 2002 Aug;55(8):60-4. No abstract available. PMID 14765452
- [Background] Lee JC, Sykes C, Saifuddin A, Connell D. Adhesive capsulitis: sonographic changes in the rotator cuff interval with arthroscopic correlation. Skeletal Radiol. 2005 Sep;34(9):522-7. doi: 10.1007/s00256-005-0957-0. Epub 2005 Jul 6. PMID 15999280
- [Background] Murnaghan JP. Frozen Shoulder, in Rockwood CA Jr, Matsen FA III (eds): The Shoulder. Philadelphia: WB Saunders, 1990, pp 837-62.
- [Background] Neviaser TJ. Arthroscopy of the shoulder. Orthop Clin North Am. 1987 Jul;18(3):361-72. PMID 3441361
- [Background] Papatheodorou A, Ellinas P, Takis F, Tsanis A, Maris I, Batakis N. US of the shoulder: rotator cuff and non-rotator cuff disorders. Radiographics. 2006 Jan-Feb;26(1):e23. doi: 10.1148/rg.e23. PMID 16352733
- [Background] Shaffer B, Tibone JE, Kerlan RK. Frozen shoulder. A long-term follow-up. J Bone Joint Surg Am. 1992 Jun;74(5):738-46. PMID 1624489
- [Background] Terslev L, Torp-Pedersen S, Qvistgaard E, Bliddal H. Spectral Doppler and resistive index. A promising tool in ultrasonographic evaluation of inflammation in rheumatoid arthritis. Acta Radiol. 2003 Nov;44(6):645-52. doi: 10.1080/02841850312331287759. PMID 14616209
- [Background] Terslev L, Torp-Pedersen S, Qvistgaard E, Danneskiold-Samsoe B, Bliddal H. Estimation of inflammation by Doppler ultrasound: quantitative changes after intra-articular treatment in rheumatoid arthritis. Ann Rheum Dis. 2003 Nov;62(11):1049-53. doi: 10.1136/ard.62.11.1049. PMID 14583566
- [Background] Warner JJ. Frozen Shoulder: Diagnosis and Management. J Am Acad Orthop Surg. 1997 May;5(3):130-140. doi: 10.5435/00124635-199705000-00002. PMID 10797215